CLINICAL TRIAL: NCT05450536
Title: Self-Advocacy at the University Level: Teaching Students With Autism Spectrum Disorder to Advocate for Their Needs
Brief Title: Self-Advocacy Training for Autistic College Students at a Public University
Acronym: ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mark Tapia, Principal Investigator, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Self-Advocacy ASD
Record Dates: First submitted 2022-07-01; First posted 2022-07-08 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Self-Advocacy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autism College Students (Other): Single subject design means subjects are their own control.
  Interventions: Other: Video Model and Role Play

INTERVENTIONS:
Other: Video Model and Role Play — Video clips and role-play will be utilized to teach self-advocacy skills to autistic college students.

SUMMARY:
Cases in autism spectrum disorder (ASD) have dramatically risen over the past 30 years, with the current rate of 1 in every 44 (Maenner et al., 2021) children born with the condition. Much emphasis rests on the need for various interventions, practices, and therapies during childhood to improve quality of life and success across a variety of settings. Nonetheless, as they age, all children advance through the education system and eventually leave the school system. Consequently, it should not be surprising that these children must grow up and face realities after high school. For some, this may include residential placements, living at home with family members, or working part or full time. For others, this comes in the form of postsecondary education. However, many individuals with autism might not be prepared to handle the requirements future education entails. As stated in articles by Chiang et al. (2012) and Blackorby and Wagner (1996), persons with disabilities, regardless of type, do not have successful transitions after high school compared to individuals without disabilities-even with having access to many resources in school and the community. Barriers, therefore, exist that prevent successful outcomes for students with autism attending college and obtaining a postsecondary degree. Thus, there is a need to identify strategies that can be effective in assisting autistic adults in postsecondary education to succeed, both academically and socially.

DETAILED DESCRIPTION:
This study will utilize a concurrent multiple baseline design across participants with an embedded ABCDE design (or more specifically, an ABACADAE design). These components will be the four scenarios teaching self-advocacy skills based primarily on recognition of one's wants and needs and personal decision making. The four included scenarios will be a) requesting appropriate accommodations from disability services; b) requesting additional supports or services (daily living, social, etc.) from disability services; c) presenting accommodations to a professor; and d) meeting with disability services in the event a professor is not accommodating student needs. There will also be a pre-test/post-test comparison between scores on the self-advocacy questionnaire with data displayed in the form of a bar graph that will explore all four areas of self-advocacy: recognition of wants and needs, scheduling meetings, locating services, and personal decision making.

ELIGIBILITY:
Inclusion Criteria:

* Students to be undergraduates enrolled at a university or community college
* Students must have a confirmed diagnosis of ASD (either through an official diagnosis via documentation of the disability services or proof of self-diagnosis).

Exclusion Criteria:

* Students who are not enrolled in college, do not have a confirmed diagnosis of ASD, or who already demonstrate strong self-advocacy skills will be excluded from this study.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Advocacy Skills | Through study completion, which will be up to 3 months
  Self-Advocacy Questionnaire-a 16 question survey that looks at 4 areas of self-advocacy. 4 questions per each scenario leading to the total of 16. Numerical values are not used to measure specific variables--but they are used to compare and contrast how participants answered the questionnaire at a pretest and posttest basis.

SECONDARY OUTCOMES:
Social Validity Application of the Intervention Package | At the end of the study, which on average will last up to 3 months.
  Social Validity Questionnaire will assess the accuracy of the measures this study used--i.e., video model, script, and task-analysis. This is a 6 question survey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided